CLINICAL TRIAL: NCT01530906
Title: Efficiency of rTMS in Bulimia: a Controlled Randomized Study
Brief Title: Efficiency of Repetitive Transcranial Magnetic Stimulation (rTMS) in Bulimia
Acronym: rTMS&bulimia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Saint Etienne (Other); University Hospital, Marseille (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8709; 2011-A01018-33 (Other: ID-RCB (Afssaps))
Record Dates: First submitted 2012-02-01; First posted 2012-02-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2012-02

CONDITIONS: Bulimia Nervosa
Keywords: Eating disorders; Bulimia; rTMS; Treatment
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders; Bulimia | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rTMS (Experimental): patients included in this arm will receive 10 sessions of transcranial magnetic stimulation (10 TMS sessions of 20 trains of 5s with 55s interval cross train, at a frequency of 10 Hz and 110% of motor threshold intensity of the left DLPFC).
  Fifty percent of patients will be included in this arm. During the first and last session a food challenge task will be administered before and after rTMS. Salivary cortisol level will be assessed throughout the protocol Intervention: Repetitive transcranial Magnetic Stimulation (rTMS)
  Interventions: Procedure: Repetitive transcranial Magnetic Stimulation (rTMS)
- rTMS SHAM (Placebo Comparator): Transcranial magnetic stimulation SHAM Intervention: Repetitive transcranial Magnetic Stimulation SHAM Fifty percent of patients will be included in this arm. During the first and last session a food challenge task will be administered before and after rTMS. Salivary cortisol level will be assessed throughout the protocol
  Interventions: Procedure: Repetitive transcranial Magnetic Stimulation SHAM

INTERVENTIONS:
Procedure: Repetitive transcranial Magnetic Stimulation (rTMS) — 10 TMS sessions of 20 trains of 5s with 55s interval cross train, at a frequency of 10 Hz and 110% of motor threshold intensity of the left DLPFC.
  Other Names: Magstim rapid2; Reference 3576-23-05
  Arms: rTMS
Procedure: Repetitive transcranial Magnetic Stimulation SHAM — Sham treatment will be performed with a placebo coil. The same coil as coil used for rTMS, but it does not deliver magnetic field.
  Other Names: Magstim Company
  Arms: rTMS SHAM

SUMMARY:
Bulimia nervosa is defined by recurrent episodes of binge eating followed by compensatory behaviors (such as induced vomiting) to prevent weight gain. It is a common and serious disease for which current treatment strategies have to be improved.

The aim of this study is to assess whether a transcranial magnetic stimulation reduces bulimic symptoms in a short term.

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a noninvasive outpatient technique of brain stimulation, based on the delivery of the localized magnetic field. It is now widely used a in a variety of neurological and psychiatric disorders.

Several clinical and pathophysiological studies suggest efficacy of rTMS on the reduction of craving and/or addictive behavior in various addictions such as alcoholism, smocking or cocaine. Because of the addictive design of the BN, the effect of one session of rTMS on food craving has been tested.

These studies show that stimulation of left dorsolateral prefrontal cortex (DPLPFC) under high frequency decreases craving food. In addition, in a healthy subject, studies show that rTMS appear to alter neuropsychological functions very involved in physiopathology of bulimia. To date, the investigators do not know if rTMS cold be a useful treatment in the treatment of bulimia. But in the light of these data, the investigators hypothesize that a program of rtMS may have a therapeutic effect and therefore an interest for the treatment of bulimia.

The objective of this project is to assess whether a program of repetitive transcranial magnetic stimulation (rTMS) under high frequency at the left DLPFC reduces bulimic symptoms in the short term.

This is a french multicenter study (Montpellier, Marseille, Saint Etienne), randomized, single blind, two arm, in addition of a treatment already validated (prescription of selective inhibitors of serotonin reuptake inhibitors (SSRIs)). The two arms are : one arm with SSRI + rTMS and an arm with SSRI + sham rTMS (placebo), 30 patients per group will be recruited.

The methodology includes:

1. an initial clinical and neuropsychological assessment.
2. 10 TMS sessions of 20 trains of 5s with 55s interval cross train, at a frequency of 10 Hz and 110% of motor threshold intensity of the left DLPFC. Fifty percent of patients will have a real stimulation and and the other fifty percent a sham stimulation. Subjects will be randomized to one or other of the two groups. During the first and last session a food challenge task will be administered before and after rTMS. Salivary cortisol level will be assessed throughout the protocol.
3. the final clinical and neuropsychological assessment at 1 month (15 days minimum after the last Session of rTMS).

The primary endpoint will focus on the number of binge within 15 days after the last session of rTMS.

If the investigators hypothesis is confirmed the investigators will highlight a new therapeutic modality in the treatment of bulimia. The secondary objectives will permit a better understanding of the pathophysiology of the disorder and ways of possible therapeutic actions of rTMS

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of bulimia nervosa (DSM IV)
* Women (18-40 years old)
* right-handed
* treated by fluoxetine (60mg/j) or escitalopram (30mg/j) for at least 3 weeks.
* use effective contraceptive measures

Exclusion criteria:

* Current anorexia as DSM IV criteria
* Current psychiatric disorder unstabilized
* Taking corticosteroid
* History of seizures or epilepsy
* History of head trauma, cerebral pathology
* Serious physical illness unstabilized
* Prior use of the TMS
* pregnancy or breastfeeding
* Somatic disease may affect cognitive abilities and brain structures
* Loss of personal capacity resulting in state protection
* Deprivation of liberty by judicial or administrative decision
* Patients with pacemakers, defibrillator, neuro stimulator implanted.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-01; Primary Completion 2015-03 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Efficiency of rTMS in bulimia | At J0 and J45 (maximum of 45 days between the inclusion visit and the final visit)
  The objective of this project is to assess whether a program of repetitive transcranial magnetic stimulation (rTMS) under high frequency at the left DLPFC reduces bulimic symptoms in the short term. To do this we will count the number of binge during the 15 days following the last session of rTMS.

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Guillaume, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

REFERENCES:
- [Result] Van den Eynde F, Guillaume S, Broadbent H, Campbell IC, Schmidt U. Repetitive transcranial magnetic stimulation in anorexia nervosa: a pilot study. Eur Psychiatry. 2013 Feb;28(2):98-101. doi: 10.1016/j.eurpsy.2011.06.002. Epub 2011 Aug 30. PMID 21880470
- [Result] Van den Eynde F, Broadbent H, Guillaume S, Claudino A, Campbell IC, Schmidt U. Handedness, repetitive transcranial magnetic stimulation and bulimic disorders. Eur Psychiatry. 2012 May;27(4):290-3. doi: 10.1016/j.eurpsy.2010.08.015. Epub 2010 Nov 9. PMID 21067901
- [Derived] Guillaume S, Gay A, Jaussent I, Sigaud T, Billard S, Attal J, Seneque M, Galusca B, Thiebaut S, Massoubre C, Courtet P. Improving decision-making and cognitive impulse control in bulimia nervosa by rTMS: An ancillary randomized controlled study. Int J Eat Disord. 2018 Sep;51(9):1103-1106. doi: 10.1002/eat.22942. Epub 2018 Sep 21. PMID 30240526